CLINICAL TRIAL: NCT00230334
Title: Phase II Study of Gleevec (Imatinib Mesylate) in Patients With Idiopathic Hypereosinophilic Syndrome (HES)
Brief Title: Phase II Gleevec Idiopathic Hypereosinophilic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated by PI due to insufficient accrual
Sponsor: Steven E. Coutre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Professor of Medicine (Hematology) at the Stanford University Medical Center, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 79112 (old system); HEMMPD0001 (Other: OnCore)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Eosinophilia; Hypereosinophilic Syndrome
MeSH Terms: conditions — Eosinophilia; Hypereosinophilic Syndrome | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gleevec

SUMMARY:
The purpose of the trial is to determine the safety and efficacy of Gleevec" in idiopathic hypereosinophilic syndrome (HES) and to characterize the molecular basis for the therapeutic benefit of Gleevec" in HES.

ELIGIBILITY:
Inclusion Criteria:- At study entry, absolute peripheral blood eosinophil count greater than upper limit of normal at the laboratory where the analysis is performed.

* Patients must have symptomatic disease, e.g. signs or symptoms of organ involvement related to eosinophilia. Examples include pulmonary, cardiac, GI, or central nervous system disease, hepatomegaly, splenomegaly, or skin disease.
* BCR-ABL-negative by PCR.
* Patients are imatinib-naive.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow capsules.
 Exclusion Criteria:- Pregnant or nursing women. Patients of childbearing potential must have a negative pregnancy test prior to initiation of study drug. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control during the study and for 3 months following discontinuation of study drug.
* Serum creatinine >2.0.
* Total serum bilirubin >2.0 mg/dl. AST(SGOT) and ALT (SGPT) more than 2.5 x the upper limit of normal range (ULN) at the laboratory where the analyses is performed.
* Presence of clonal T-lymphocyte population by PCR or southern blotting.
* ECOG Performance Status Score > or = to 3.
* Busulfan within 6 weeks of starting treatment.
* IFN-a within 14 days of starting treatment.
* Low dose cytosine-arabinoside or vincristine within 14 days of starting treatment.
* Hydroxyurea within 1 day of starting treatment.
* Prednisone or other immunosuppressives (e.g. azathioprine, cyclosporine-A) within 14 days of starting treatment.
* AML/ALL-type induction chemotherapy within 4 weeks of starting treatment
* Persistent peripheral blood count toxicity of grade 2 or higher after receiving AML/ALL-type induction chemotherapy.
* Treatment with other investigational agents within 28 days of starting treatment.
* History of non-compliance to medical regimens.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (Grade 3 / 4 New York Heart Association Criteria), unstable angina pectoris or cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of HIV-positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-06-12 (Actual); Primary Completion 2006-12-29 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the hematologic response rate of imatinib in patients with HES.

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Coutre, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States